CLINICAL TRIAL: NCT04591444
Title: Efficacy of a Fluoride Varnish and a Glass Ionomer Sealant on Cervical Dentin Hypersensitivity: A Randomized Clinical Trial
Brief Title: Fluoride Varnish X Glass Ionomer Sealant on Cervical Dentin Hypersensitivity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fausto Medeiros Mendes, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HDFOUSP
Record Dates: First submitted 2020-10-11; First posted 2020-10-19 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Dentin Hypersensitivity; Dentin Sensitivity
Keywords: Dentin hypersensitivity; Dentin sensitivity; Hypersensitivity; Fluorides; Sodium fluoride; Glass ionomer sealant; Desensitizing treatment; Glass ionomer cement
MeSH Terms: conditions — Dentin Sensitivity; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: The present study is a parallel, randomized, triple blind clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ClinproTM White Varnish (Active Comparator): Application of ClinproTM White Varnish containing sodium fluoride (5%) and Tricalcium phosphate (TCP).
  A technology that allows calcium and phosphate ions to coexist with fluoride ions separately, forming a more resistant mineral on the tooth surface (3M ESPE Clinpro White Varnish; 3M ESPE Clinpro 5000).
  Interventions: Drug: Fluoride Varnish
- ClinproTM XT Varnish (Active Comparator): Application of ClinproTM XT Varnish, a resin-modified glass ionomer sealant.
  Creates a protective layer on exposed dentin, which is durable and has the ability to release fluoride, calcium and phosphate into the surroundings. (3M ESPE Clinpro XT Varnish).
  Interventions: Drug: Glass Ionomer Sealant
- Placebo Group (Placebo Comparator): Participants who were part of the placebo group continuously used only the conventional toothpaste provided in the oral hygiene kit during the initial four weeks of the research and received a simulated treatment.
  Interventions: Other: Placebo Group

INTERVENTIONS:
Drug: Fluoride Varnish — Following the manufacturer's recommendations, it was not necessary to moisten or dry the treated surface beforehand or afterwards. The product was dispensed and manipulated for 15 s until a homogeneous mixture was obtained, applied with a micro brush, flowing into interproximal areas, and quickly adhering to the tooth surface in the presence of saliva.
  Other Names: ClinproTM White Varnish
  Arms: ClinproTM White Varnish
Drug: Glass Ionomer Sealant — Following the manufacturer's recommendations, prophylaxis and prior drying of the treated surface was carried out, the product was also dispensed and manipulated for 15 s until a homogeneous mixture was obtained, applied with a micro brush and light-cured for 20 s.
  Other Names: ClinproTM XT Varnish; Resin-modified Glass Ionomer Sealant
  Arms: ClinproTM XT Varnish
Other: Placebo Group — 4 weeks after the simulation of the treatment application, participants in the placebo group received DH treatment with the product that had the best effect in the first 4 weeks.
  Arms: Placebo Group

SUMMARY:
Dentin hypersensitivity (DH) can be defined as acute, short-duration pain from open dentin tubules in exposed dentin. The symptom of DH is subjective and varies from patient to patient and may present as mild discomfort or as a high-intensity pain, which can affect the individual's quality of life, interfering with their eating and hygiene habits. One approach to treatment would be the use of agents that chemically desensitize sensory nerves, blocking the transmission of nerve stimuli to the central nervous system.

The effectiveness of desensitizing treatments is influenced by several factors present in the oral cavity, which can contribute to a greater effect of these agents but can also be responsible for removing them from the dental surface. To date, studies have been carried out in the short term, not exceeding an average period of 12 weeks, so there is no consensus on the technique or agent that will guarantee the most effective and lasting effect against DH, not even the ideal period for reapplication. Thus, more studies are needed to assess the clinical behavior of desensitizing products on the market, especially the most recent releases. Therefore, the aim of this study was to clinically compare the effectiveness of different office treatments for DH, being ClinproTM White Varnish, ClinproTM XT Varnish, and a control group (placebo) through pain assessment with the Visual Analog Scale (VAS), after stimulation with air from the triple syringe.

DETAILED DESCRIPTION:
This study compares the effectiveness of two in-office treatment for dentin hypersensitivity: G1:ClinproTM White Varnish, G2:ClinproTM XT Varnish, and a G3:placebo (where the application of a product was only simulated). Recruitment of the 121 volunteers were based on their self-reported complaint of dentin hypersensitivity, which confirmed with the use of an air blast from a triple syringe. Then, he/she showed in the VAS scale (which varies from 0=no pain to 10=the worst pain possible) the value that best describes the pain sensation. The subjects that present at least one tooth with a value of 4 and above in the VAS scale (if more than one hypersensitive tooth was present, the mean VAS values obtained were used, for each patient) was randomly allocated into the experimental groups. Two weeks before the study started, the volunteers went through a wash out period, where they used only the oral hygiene products donated by the researchers, which were used up to the end of the study. The in-office treatments were performed after prophylaxis, according to the manufacturer´s instructions, by one trained researcher, which was blind to the treatments. DH evaluation was performed 15 min after the application of the treatments, by a different researcher, which also blind to the treatment, and which used the same methodology described early for the detection of initial pain. The volunteers were recalled for the DH evaluation after one and four weeks of the treatments. DH evaluation was also performed after 12 and 24 weeks of the treatments, except in the placebo group, which received the proper DH treatment after the first four weeks of the study. Data was analyzed with the appropriate statistical methods (α=0.05).

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years old;
* Presented good general health;
* Presented at least one tooth with DH reported in the cervical region, which has a graded sensitivity of 4 or more on the VAS scale.

Exclusion Criteria:

* Presented active caries lesions or with defective restorations in the tooth to be analyzed;
* Presented enough dentin loss that required restorative treatment or periodontal surgery;
* Volunteers who underwent any professional desensitizing treatment in the last 6 months;
* Volunteers who used desensitizing pastes in the 3 months;
* Volunteers who were using anti-inflammatory or analgesic drugs at the time of recruitment;
* Volunteers were are pregnant or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Change in the dentin hypersensitivity | 4 weeks
  The evaluation was performed with the use of Visual Analog Scale (VAS). The volunteers pointed out on the VAS (ranging from 0=no pain to 10=worst possible pain) the whole number, which best described his perception of pain at the moment.
  The primary outcome was the difference between the Visual Analog Scale values obtained in the baseline and 4 weeks after the treatment.

SECONDARY OUTCOMES:
Dentin hypersensitivity | baseline, 15 minutes after the treatments, 1 week and 4 weeks.
  This secondary outcome was the Visual Analog Scale (VAS) score related to dentin hypersensitivity. The volunteers pointed out on the VAS (ranging from 0=no pain to 10=worst possible pain) the whole number, which best described his perception of pain at the moment.
  Visual Analog Scale was applied before the treatment (baseline), 15 minutes after the procedures, one week, and 4 weeks after treatments to measure the changes in dentin hypersensitivity.
Change in the dentin hypersensitivity | 3 months and 6 months
  The evaluation was performed with the use of Visual Analog Scale (VAS). The volunteers pointed out on the VAS (ranging from 0=no pain to 10=worst possible pain) the whole number, which best described his perception of pain at the moment.
  This secondary outcome was the difference between the Visual Analog Scale values obtained in the baseline and 3 and 6 months after the treatment (Long-term differences in the VAS values).

CONTACTS AND LOCATIONS:
Overall Officials: Taís Scaramucci Forlin, Assistant Professor, Principal Investigator — University of Sao Paulo
Locations (1):
- School of Dentistry, University of Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Machado AC, Maximiano V, Yoshida ML, Freitas JG, Mendes FM, Aranha ACC, Scaramucci T. Efficacy of a calcium-phosphate/fluoride varnish and ionomeric sealant on cervical dentin hypersensitivity: A randomized, double-blind, placebo-controlled clinical study. J Oral Rehabil. 2022 Jan;49(1):62-70. doi: 10.1111/joor.13270. Epub 2021 Nov 2. PMID 34676918